CLINICAL TRIAL: NCT01064414
Title: A Randomized, Double-Blind, Placebo-Controlled, 3-Arm, Parallel-Group, 26-Week, Multicenter Study With a 26-Week Extension, to Evaluate the Efficacy, Safety and Tolerability of Canagliflozin in the Treatment of Subjects With Type 2 Diabetes Mellitus Who Have Moderate Renal Impairment
Brief Title: An Efficacy, Safety, and Tolerability Study of Canagliflozin in Patients With Type 2 Diabetes Mellitus Who Have Moderate Renal Impairment
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CR017008; 28431754DIA3004 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2010-02-04; First posted 2010-02-08 (Estimated); Results first posted 2013-05-27 (Estimated); Last update posted 2013-08-14 (Estimated); Status verified 2013-08

CONDITIONS: Diabetes Mellitus, Type 2; Renal Insufficiency
Keywords: Canagliflozin; JNJ 28431754; Placebo; Sodium-Glucose Transporter 2; hemoglobin A1c protein, Blood Glucose; reduced kidney function, Type 2 diabetes mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Renal Insufficiency | interventions — Canagliflozin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Canagliflozin 100 mg (Experimental): Each patient will receive 100 mg of canagliflozin once daily for 52 weeks.
  Interventions: Drug: Canagliflozin
- Canagliflozin 300 mg (Experimental): Each patient will receive 300 mg of canagliflozin once daily for 52 weeks.
  Interventions: Drug: Canagliflozin
- Placebo (Placebo Comparator): Each patient will receive matching placebo once daily for 52 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Canagliflozin — One 100 mg or 300 mg over-encapsulated tablet orally (by mouth) once daily for 52 weeks in addition to the patient's AHA regimen used in accordance with local prescribing information
  Arms: Canagliflozin 100 mg; Canagliflozin 300 mg
Drug: Placebo — One matching placebo capsule orally once daily for 52 weeks in addition to the patient's AHA regimen used in accordance with local prescribing information
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of 2 different doses of canagliflozin compared with placebo in patients with type 2 diabetes mellitus who have reduced kidney function.

DETAILED DESCRIPTION:
This is a randomized (study drug assigned by chance), double blind (neither the patient or the study doctor will know the name of the assigned treatment), parallel-group, 3-arm (patients will be assigned to 1 of 3 treatment groups) multicenter study to determine the efficacy, safety, and tolerability of 2 different doses of canagliflozin (100 mg and 300 mg) compared to placebo (a pill that looks like all the other treatments but has no real medicine) in patients with type 2 diabetes mellitus (T2DM) who have renal impairment (reduced kidney function) and who are not achieving an adequate response from current therapy to control their diabetes. Canagliflozin (also referred to as JNJ-28431754) is a drug that is being tested to see if it may be useful in treating patients diagnosed with T2DM. Approximately 240 patients will participate in the study for approximately 63 to 72 weeks, depending on the length of the pretreatment phase. The study will consist of a pretreatment phase, a 52 week double blind treatment phase, and a posttreatment phase. During the pretreatment phase, screening evaluations will be performed to see if patients meet the entry criteria for the study. In addition, routine clinical procedures will be performed (physical examination, vital signs measurements, and an electrocardiogram [ECG]), a blood and urine sample will be collected for routine clinical laboratory tests, and all antihyperglycemic therapy taken by patients will be reviewed. Patients who meet entrance criteria for the study and who currently take a stable antihyperglycemic agent (AHA) regimen according to the local prescribing information will be eligible for inclusion in the study. Patients who meet entrance criteria for the study but who are not taking a stable AHA regimen according to the local prescribing information will enter an AHA adjustment period that may last for up to 12 weeks. Patients will receive once daily treatment with study drug in addition to their current stable diabetes regimen (eg, diet, exercise, and medication therapy). Patients will continue to take their assigned treatment for 52 weeks (includes a 26-week core double-blind treatment period and a 26-week extension double-blind treatment period). During the study, if a patient's blood sugar remains high despite treatment with study drug in combination with their other antidiabetic agents, the study physician will modify the patient's treatment. If patients take insulin and experience low blood sugar (hypoglycemia), the dose of insulin may be modified. During the study, patients will be monitored for safety by review of adverse events, results from safety laboratory tests (including chemistry, hematology, and urinalysis), ECGs, vital signs measurements, body weight, physical examinations, self-monitored blood glucose, and collection of potential hypoglycemic episodes reported by patients on diary cards. The safety of patients in this study will also be monitored by a company internal Medical Safety Review Committee (MSRC). An Independent Data Monitoring Committee (IDMC) will evaluate cardiovascular (CV) events that are reported across the entire clinical development program for canagliflozin. Patients who complete the Week 52 visit or who discontinue treatment early and are withdrawn from the study will have end-of-study evaluations performed and a follow-up telephone interview conducted by study personnel approximately 30 days (but no more than 42 days) after the last dose of study drug to collect any serious adverse events that occurred since their last study visit. The primary outcome measures in the study are to assess the effect of canagliflozin relative to placebo on hemoglobin A1c (HbA1c, a blood test used to measure the control of diabetes) after 26 weeks of treatment and to assess the safety and tolerability of canagliflozin from time of signed informed consent to study end (includes up to 30 days following the last dose of study drug). All patients will take a single-blind placebo capsule once daily for 2 weeks before randomization to double-blind study drug. After randomization, patients will take one capsule of canagliflozin (either 100 mg or 300 mg) or matching placebo orally (by mouth) with liquid once daily for 52 weeks before the first meal each day except on days when fasting or pharmacokinetic blood samples are collected in which case study drug will be taken after the visit immediately before the patient's next meal.

ELIGIBILITY:
Inclusion Criteria:

* Patients with T2DM not on an AHA or on any AHA in monotherapy or combination therapy (including oral or non oral agents)
* Patients with reduced kidney function

Exclusion Criteria:

* History of diabetic ketoacidosis, type 1 diabetes mellitus (T1DM), pancreas or beta cell transplantation, or diabetes secondary to pancreatitis or pancreatectomy
* Have proliferative diabetic retinopathy for which treatment is planned during the course of the study
* Kidney disease that required treatment with immunosuppressive therapy, history of dialysis or kidney transplant, presence of nephrotic syndrome (eg, severe proteinuria with hypoalbuminemia and/or edema), or inflammatory kidney disease
* Receiving anti hypertensive or anti-hyperlipidemic therapy not on a stable regimen
* History of a severe hypoglycemic episode within 6 months before screening

Min Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 272 (Actual)
Dates: Start 2010-06; Primary Completion 2011-12 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC C. Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (106):
- United States (26):
  - Concord, California
  - Fountain Valley, California
  - San Diego, California
  - Denver, Colorado
  - Pembroke Pines, Florida
  - Tampa, Florida
  - West Palm Beach, Florida
  - Augusta, Georgia
  - Nampa, Idaho
  - Baton Rouge, Louisiana
  - Jackson, Mississippi
  - Picayune, Mississippi
  - Chesterfield, Missouri
  - Las Vegas, Nevada
  - Albuquerque, New Mexico
  - Durham, North Carolina
  - Canal Fulton, Ohio
  - Cincinnati, Ohio
  - Columbus, Ohio
  - Zanesville, Ohio
  - Oklahoma City, Oklahoma
  - Meridian, Pennsylvania
  - Pittsburgh, Pennsylvania
  - North Charleston, South Carolina
  - Salt Lake City, Utah
  - Fairfax, Virginia
- Australia (4):
  - Camperdown
  - Gosford
  - Parkville
  - Reservoir
- Belgium (6):
  - Aalst
  - Bonheiden
  - Brussels
  - Liège
  - Sint-Niklaas
  - Turnhout
- São Paulo, Brazil
- Canada (10):
  - Vancouver, British Columbia
  - Victoria, British Columbia
  - Antigonish, Nova Scotia
  - Sydney, Nova Scotia
  - Hamilton, Ontario
  - London, Ontario
  - Smiths Falls, Ontario
  - Thornhill, Ontario
  - Montreal, Quebec
  - Calgary
- France (7):
  - Corbeil-Essonnes
  - La Rochelle Cedex 1 Poitou-Cha
  - Le Creusot
  - Nantes
  - Pierre-Bénite
  - Vandœuvre-lès-Nancy
  - Vénissieux
- Germany (9):
  - Dormagen
  - Dortmund
  - Dresden
  - Einbeck
  - Freiburg im Breisgau
  - Kassel
  - München
  - Schkeuditz
  - Würzburg
- India (3):
  - Aurangabad
  - Madurai
  - Pune
- Latvia (3):
  - Daugavpils
  - Ogre
  - Riga
- Malaysia (4):
  - Jalan Cheras N/A
  - Kajang
  - Kuala Lumpur
  - Pulau Pinang
- Mexico (4):
  - Aguascalientes
  - Culiacán
  - Morelia
  - Zapopan
- New Zealand (4):
  - Auckland
  - Christchurch
  - Dunedin Nz
  - Nz
- Poland (3):
  - Lublin
  - Warsaw
  - Łask
- Romania (2):
  - Bucharest
  - Târgovişte
- Russia (9):
  - Chelyabinsk
  - Kirov
  - Kursk
  - Moscow
  - Nizhny Novgorod
  - Petrozavodsk
  - Rostov-on-Don
  - Saint Petersburg
  - Yaroslavl
- South Africa (3):
  - Parow, Cape Town
  - Pretoria
  - Somerset West
- South Korea (2):
  - Seognam-Si, Kyungki-Do
  - Seoul
- Spain (6):
  - Barcelona
  - Ciudad Real
  - Madrid
  - San Sebastián de los Reyes
  - Santa Cruz de Tenerife
  - Valencia

REFERENCES:
- [Derived] Watts NB, Bilezikian JP, Usiskin K, Edwards R, Desai M, Law G, Meininger G. Effects of Canagliflozin on Fracture Risk in Patients With Type 2 Diabetes Mellitus. J Clin Endocrinol Metab. 2016 Jan;101(1):157-66. doi: 10.1210/jc.2015-3167. Epub 2015 Nov 18. PMID 26580237
- [Derived] Weir MR, Kline I, Xie J, Edwards R, Usiskin K. Effect of canagliflozin on serum electrolytes in patients with type 2 diabetes in relation to estimated glomerular filtration rate (eGFR). Curr Med Res Opin. 2014 Sep;30(9):1759-68. doi: 10.1185/03007995.2014.919907. Epub 2014 May 22. PMID 24786834
- [Derived] Nyirjesy P, Sobel JD, Fung A, Mayer C, Capuano G, Ways K, Usiskin K. Genital mycotic infections with canagliflozin, a sodium glucose co-transporter 2 inhibitor, in patients with type 2 diabetes mellitus: a pooled analysis of clinical studies. Curr Med Res Opin. 2014 Jun;30(6):1109-19. doi: 10.1185/03007995.2014.890925. Epub 2014 Feb 21. PMID 24517339

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study evaluated the efficacy and safety of canagliflozin in patients with type 2 diabetes mellitus and moderate renal impairment. The study was conducted between 02 March 2010 and 19 January 2012 and recruited patients from 89 study centers located in 19 countries worldwide.
Pre-assignment Details: 272 patients were randomly allocated to the 3 treatment arms. 269 patients received at least 1 dose of study drug and were included in the modified intent-to-treat (mITT) analysis set and safety analysis set. Participant flow is presented in two parts: for Baseline to Week 26 as "Core Period", and for Week 26 to Week 52 as "Extension Period".
Groups:
- Placebo: Each patient received matching placebo once daily for 52 weeks. Data are presented for Baseline to Week 26 (Core Period) and for Week 26 to 52 (Extension Period).
- Canagliflozin 100 mg: Each patient received 100 mg of canagliflozin once daily for 52 weeks. Data are presented for Baseline to Week 26 (Core Period) and for Week 26 to 52 (Extension Period).
- Canagliflozin 300 mg: Each patient received 300 mg of canagliflozin once daily for 52 weeks.Data are presented for Baseline to Week 26 (Core Period) and for Week 26 to 52 (Extension Period).
Period: Core Period: Baseline to Week 26
Arm/Group | Placebo | Canagliflozin 100 mg | Canagliflozin 300 mg
Started | 90 | 90 | 89
Completed | 77 | 75 | 82
Not Completed | 13 | 15 | 7
Not completed — Adverse Event | 4 | 4 | 2
Not completed — Death | 0 | 1 | 0
Not completed — Protocol Violation | 1 | 0 | 1
Not completed — Withdrawal by Subject | 4 | 2 | 2
Not completed — Noncompliance with study drug | 0 | 1 | 0
Not completed — Other | 4 | 7 | 2
Period: Extension Period: Week 26 to Week 52
Arm/Group | Placebo | Canagliflozin 100 mg | Canagliflozin 300 mg
Started | 76 (1 pt completed core but did not enter ext. Reason: other (not specified).) | 72 (3 pts completed core but did not enter ext. Reason: other (not specified) (3).) | 81 (1 pt completed core but did not enter ext. Reason: other (not specified).)
Completed | 64 | 67 | 76
Not Completed | 12 | 5 | 5
Not completed — Adverse Event | 2 | 1 | 2
Not completed — Death | 0 | 1 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0
Not completed — Physician Decision | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 1
Not completed — Noncompliance with study drug | 1 | 0 | 0
Not completed — Protocol Violation | 1 | 1 | 1
Not completed — Other | 5 | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Placebo: Each patient received matching placebo once daily for 52 weeks.
- Canagliflozin 100 mg: Each patient received 100 mg of canagliflozin once daily for 52 weeks.
- Canagliflozin 300 mg: Each patient received 300 mg of canagliflozin once daily for 52 weeks.
- Total: Total of all reporting groups
Arm/Group | Placebo | Canagliflozin 100 mg | Canagliflozin 300 mg | Total
Number analyzed (Participants) | 90 | 90 | 89 | 269
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 27 | 24 | 32 | 83
  >=65 years | 63 | 66 | 57 | 186
Age Continuous [Mean (Standard Deviation); unit: years] | 68.2 (8.4) | 69.5 (8.2) | 67.9 (8.24) | 68.5 (8.28)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 32 | 41 | 106
  Male | 57 | 58 | 48 | 163
Region of Enrollment [Number; unit: participants]
  AUSTRALIA | 3 | 6 | 5 | 14
  BELGIUM | 5 | 1 | 6 | 12
  BRAZIL | 4 | 4 | 5 | 13
  CANADA | 7 | 11 | 3 | 21
  FRANCE | 7 | 5 | 4 | 16
  GERMANY | 6 | 10 | 2 | 18
  INDIA | 3 | 3 | 3 | 9
  ITALY | 4 | 1 | 1 | 6
  LATVIA | 2 | 1 | 4 | 7
  MALAYSIA | 2 | 4 | 8 | 14
  MEXICO | 0 | 2 | 2 | 4
  NEW ZEALAND | 7 | 2 | 5 | 14
  POLAND | 5 | 5 | 4 | 14
  ROMANIA | 2 | 1 | 2 | 5
  RUSSIAN FEDERATION | 10 | 11 | 9 | 30
  SOUTH AFRICA | 2 | 3 | 1 | 6
  SOUTH KOREA | 1 | 1 | 0 | 2
  SPAIN | 4 | 5 | 8 | 17
  UNITED STATES | 16 | 14 | 17 | 47

OUTCOME MEASURES:

1. Primary Outcome: Change in HbA1c From Baseline to Week 26
Description: The table below shows the least-squares (LS) mean change in HbA1c from Baseline to Week 26 for each treatment group. The statistical analyses show the treatment differences (ie, each canagliflozin group minus placebo) in the LS mean change.
Time Frame: Day 1 (Baseline) and Week 26
Population: Analysis used mITT analysis set (all randomized patients who received at least 1 dose of study drug). Last-observation-carried-forward method used for missing Week 26 values. Measurements taken pre-rescue used as last observation in patients receiving glycemic rescue therapy. Table includes only patients with both baseline and post baseline values.
Measure: Least Squares Mean (Standard Error); unit: Percent
Groups:
- Canagliflozin 100 mg: Each patient received canagliflozin 100 mg once daily for 52 weeks.
- Canagliflozin 300 mg: Each patient received canagliflozin 300 mg once daily for 52 weeks.
Arm/Group | Placebo | Canagliflozin 100 mg | Canagliflozin 300 mg
Number analyzed (Participants) | 87 | 88 | 89
Percent | -0.03 (0.090) | -0.33 (0.090) | -0.44 (0.089)
Statistical Analysis 1: Comparison: Placebo vs Canagliflozin 100 mg; Test type: Superiority or Other; p = 0.012, ANCOVA; Least-Squares Mean Difference = -0.30, 95% CI 2-sided [-0.529 to -0.066], Standard Error of Mean 0.117
Statistical Analysis 2: Comparison: Placebo vs Canagliflozin 300 mg; Test type: Superiority or Other; p < 0.001, ANCOVA; Least-Squares Mean Difference = -0.40, 95% CI 2-sided [-0.635 to -0.174], Standard Error of Mean 0.117

2. Secondary Outcome: Percentage of Patients With HbA1c <7% at Week 26
Description: The table below shows the percentage of patients with HbA1c <7% at Week 26 in each treatment group. The statistical analyses show the treatment differences (ie, each canagliflozin group minus placebo) in the percentage.
Time Frame: Week 26
Population: as for outcome 1
Measure: Number; unit: Percentage of patients
Arm/Group | Placebo | Canagliflozin 100 mg | Canagliflozin 300 mg
Number analyzed (Participants) | 87 | 88 | 89
Percentage of patients | 17.2 | 27.3 | 32.6
Statistical Analysis 1: Comparison: Placebo vs Canagliflozin 100 mg; Test type: Superiority or Other; p = 0.227, Regression, Logistic; Odds Ratio (OR) = 1.66, 95% CI 2-sided [0.73 to 3.77]
Statistical Analysis 2: Comparison: Placebo vs Canagliflozin 300 mg; Test type: Superiority or Other; p = 0.017, Regression, Logistic; Odds Ratio (OR) = 2.69, 95% CI 2-sided [1.19 to 6.04]

3. Secondary Outcome: Change in Fasting Plasma Glucose (FPG) From Baseline to Week 26
Description: The table below shows the least-squares (LS) mean change in FPG from Baseline to Week 26 for each treatment group. The statistical analyses show the treatment differences (ie, each canagliflozin group minus placebo) in the LS mean change.
Time Frame: Day 1 (Baseline) and Week 26
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo | Canagliflozin 100 mg | Canagliflozin 300 mg
Number analyzed (Participants) | 88 | 90 | 88
mg/dL | 0.49 (5.089) | -14.9 (5.089) | -11.7 (5.099)
Statistical Analysis 1: Comparison: Placebo vs Canagliflozin 100 mg; Test type: Superiority or Other; p = 0.021, ANCOVA; Least-Squares Mean Difference = -15.4, 95% CI 2-sided [-28.45 to -2.307], Standard Error of Mean 6.638
Statistical Analysis 2: Comparison: Placebo vs Canagliflozin 300 mg; Test type: Superiority or Other; p = 0.069, ANCOVA; Least-Squares Mean Difference = -12.2, 95% CI 2-sided [-25.36 to 0.962], Standard Error of Mean 6.683

ADVERSE EVENTS:
Time Frame: Adverse events data were collected for the duration of study (52 weeks).
Description: The total number of adverse events listed in the "Other (non-Serious) Adverse Events" table is based upon a cut-off of greater than or equal to 5 percent of patients experiencing the adverse event in any treatment arm.
Groups:
- Placebo: Baseline to Week 26: Each patient received matching placebo once daily for 52 weeks. Data are presented for Baseline to Week 26.
- Canagliflozin 100 mg: Baseline to Week 26: Each patient received 100 mg of canagliflozin once daily for 52 weeks. Data are presented for Baseline to Week 26.
- Canagliflozin 300 mg: Baseline to Week 26: Each patient received 300 mg of canagliflozin once daily for 52 weeks. Data are presented for Baseline to Week 26.
- Placebo: Baseline to Week 52: Each patient received matching placebo once daily for 52 weeks. Data are presented for Baseline to Week 52.
- Canagliflozin 100 mg: Baseline to Week 52: Each patient received 100 mg of canagliflozin once daily for 52 weeks. Data are presented for Baseline to Week 52.
- Canagliflozin 300 mg: Baseline to Week 52: Each patient received 300 mg of canagliflozin once daily for 52 weeks. Data are presented for Baseline to Week 52.
Arm/Group | Placebo: Baseline to Week 26 | Canagliflozin 100 mg: Baseline to Week 26 | Canagliflozin 300 mg: Baseline to Week 26 | Placebo: Baseline to Week 52 | Canagliflozin 100 mg: Baseline to Week 52 | Canagliflozin 300 mg: Baseline to Week 52
Serious Adverse Events (participants affected / at risk) | 16/90 | 10/90 | 10/89 | 24/90 | 18/90 | 21/89
Other Adverse Events (participants affected / at risk) | 27/90 | 21/90 | 33/89 | 46/90 | 46/90 | 48/89
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo: Baseline to Week 26 (N=90) | Canagliflozin 100 mg: Baseline to Week 26 (N=90) | Canagliflozin 300 mg: Baseline to Week 26 (N=89) | Placebo: Baseline to Week 52 (N=90) | Canagliflozin 100 mg: Baseline to Week 52 (N=90) | Canagliflozin 300 mg: Baseline to Week 52 (N=89)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 1 | 0 — MEDDRA 14.1 used for Week 26/MEDDRA 15.0 for Week 52
Acute coronary syndrome (Cardiac disorders) | 1 | 0 | 0 | 1 | 0 | 0 — MEDDRA 14.1 used for Week 26/MEDDRA 15.0 for Week 52
Cardiac arrest (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 1 — MEDDRA 14.1 used for Week 26/MEDDRA 15.0 for Week 52
Cardiac failure congestive (Cardiac disorders) | 1 | 0 | 1 | 1 | 0 | 2 — MEDDRA 14.1 used for Week 26/MEDDRA 15.0 for Week 52
Coronary artery disease (Cardiac disorders) | 1 | 0 | 0 | 1 | 0 | 1 — MEDDRA 14.1 used for Week 26/MEDDRA 15.0 for Week 52
Myocardial infarction (Cardiac disorders) | 1 | 0 | 0 | 2 | 0 | 2 — MEDDRA 14.1 used for Week 26/MEDDRA 15.0 for Week 52
Myocardial ischaemia (Cardiac disorders) | 0 | 1 | 0 | 1 | 1 | 0 — MEDDRA 14.1 used for Week 26/MEDDRA 15.0 for Week 52
Ventricular fibrillation (Cardiac disorders) | 1 | 0 | 0 | 1 | 0 | 0 — MEDDRA 14.1 used for Week 26/MEDDRA 15.0 for Week 52
Glaucoma (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 1 — MEDDRA 14.1 used for Week 26/MEDDRA 15.0 for Week 52
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 — MEDDRA 14.1 used for Week 26/MEDDRA 15.0 for Week 52
Bile duct stone (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 1 | 0 — MEDDRA 14.1 used for Week 26/MEDDRA 15.0 for Week 52
Appendicitis perforated (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1 — MEDDRA 14.1 used for Week 26/MEDDRA 15.0 for Week 52
Campylobacter intestinal infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 — MEDDRA 14.1 used for Week 26/MEDDRA 15.0 for Week 52. In the Week 26 study report, this event was coded as "campylobacter intestinal infection"; it was subsequently re-coded in the Week 52 study report as "campylobacter gastroenteritis".
Infected skin ulcer (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1 — MEDDRA 14.1 used for Week 26/MEDDRA 15.0 for Week 52
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0 — MEDDRA 14.1 used for Week 26/MEDDRA 15.0 for Week 52
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1 — MEDDRA 14.1 used for Week 26/MEDDRA 15.0 for Week 52
Pneumonia (Infections and infestations) | 2 | 0 | 0 | 2 | 0 | 0 — MEDDRA 14.1 used for Week 26/MEDDRA 15.0 for Week 52
Sepsis (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0 — MEDDRA 14.1 used for Week 26/MEDDRA 15.0 for Week 52
Septic shock (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0 — MEDDRA 14.1 used for Week 26/MEDDRA 15.0 for Week 52
Fibula fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1 | 0 | 0 — MEDDRA 14.1 used for Week 26/MEDDRA 15.0 for Week 52
Joint dislocation (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1 | 0 | 0 — MEDDRA 14.1 used for Week 26/MEDDRA 15.0 for Week 52
Splenic rupture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 1 — MEDDRA 14.1 used for Week 26/MEDDRA 15.0 for Week 52
Tibia fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1 | 0 | 0 — MEDDRA 14.1 used for Week 26/MEDDRA 15.0 for Week 52
Wound complication (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 1 — MEDDRA 14.1 used for Week 26/MEDDRA 15.0 for Week 52
Blood creatinine increased (Investigations) | 0 | 1 | 0 | 0 | 1 | 0 — MEDDRA 14.1 used for Week 26/MEDDRA 15.0 for Week 52
Troponin increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 1 — MEDDRA 14.1 used for Week 26/MEDDRA 15.0 for Week 52
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 1 | 0 — MEDDRA 14.1 used for Week 26/MEDDRA 15.0 for Week 52
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 1 | 1 — MEDDRA 14.1 used for Week 26/MEDDRA 15.0 for Week 52
Small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 1 | 0 — MEDDRA 14.1 used for Week 26/MEDDRA 15.0 for Week 52
Carotid artery stenosis (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 1 — MEDDRA 14.1 used for Week 26/MEDDRA 15.0 for Week 52
Transient ischaemic attack (Nervous system disorders) | 1 | 1 | 0 | 1 | 1 | 0 — MEDDRA 14.1 used for Week 26/MEDDRA 15.0 for Week 52
Bladder neck obstruction (Renal and urinary disorders) | 1 | 0 | 0 | 1 | 0 | 0 — MEDDRA 14.1 used for Week 26/MEDDRA 15.0 for Week 52
Renal artery stenosis (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 1 | 0 — MEDDRA 14.1 used for Week 26/MEDDRA 15.0 for Week 52
Renal failure (Renal and urinary disorders) | 1 | 0 | 0 | 2 | 0 | 0 — MEDDRA 14.1 used for Week 26/MEDDRA 15.0 for Week 52
Renal failure acute (Renal and urinary disorders) | 0 | 1 | 1 | 1 | 1 | 1 — MEDDRA 14.1 used for Week 26/MEDDRA 15.0 for Week 52
Renal impairment (Renal and urinary disorders) | 1 | 0 | 1 | 1 | 0 | 1 — MEDDRA 14.1 used for Week 26/MEDDRA 15.0 for Week 52
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 1 | 0 — MEDDRA 14.1 used for Week 26/MEDDRA 15.0 for Week 52
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 — MEDDRA 14.1 used for Week 26/MEDDRA 15.0 for Week 52
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 1 — MEDDRA 14.1 used for Week 26/MEDDRA 15.0 for Week 52
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 0 | 0 — MEDDRA 14.1 used for Week 26/MEDDRA 15.0 for Week 52
Arteritis (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 1 — MEDDRA 14.1 used for Week 26/MEDDRA 15.0 for Week 52
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 1 | 1 | 0 | 1 — MEDDRA 14.1 used for Week 26/MEDDRA 15.0 for Week 52
Femoral arterial stenosis (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 1 — MEDDRA 14.1 used for Week 26/MEDDRA 15.0 for Week 52
Hypertension (Vascular disorders) | 1 | 0 | 0 | 1 | 0 | 0 — MEDDRA 14.1 used for Week 26/MEDDRA 15.0 for Week 52
Hypotension (Vascular disorders) | 1 | 0 | 0 | 1 | 0 | 0 — MEDDRA 14.1 used for Week 26/MEDDRA 15.0 for Week 52
Coronary artery insufficiency (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 — MEDDRA 14.1 used for Week 26/MEDDRA 15.0 for Week 52
Cor pulmonale (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 — MEDDRA 14.1 used for Week 26/MEDDRA 15.0 for Week 52
Cardiac failure acute (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 — MEDDRA 14.1 used for Week 26/MEDDRA 15.0 for Week 52
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 1 | 1 | 0 — MEDDRA 14.1 used for Week 26/MEDDRA 15.0 for Week 52
Angina pectoris (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 — MEDDRA 14.1 used for Week 26/MEDDRA 15.0 for Week 52
Angina unstable (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 — MEDDRA 14.1 used for Week 26/MEDDRA 15.0 for Week 52
Atrial fibrilation (Cardiac disorders) | 0 | 0 | 0 | 0 | 2 | 0 — MEDDRA 14.1 used for Week 26/MEDDRA 15.0 for Week 52
Cataract (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 — MEDDRA 14.1 used for Week 26/MEDDRA 15.0 for Week 52
Intestinal perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 — MEDDRA 14.1 used for Week 26/MEDDRA 15.0 for Week 52
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 — MEDDRA 14.1 used for Week 26/MEDDRA 15.0 for Week 52
Oedema peripheral (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 — MEDDRA 14.1 used for Week 26/MEDDRA 15.0 for Week 52
Appendicitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 — MEDDRA 14.1 used for Week 26/MEDDRA 15.0 for Week 52
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 — MEDDRA 14.1 used for Week 26/MEDDRA 15.0 for Week 52
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 — MEDDRA 14.1 used for Week 26/MEDDRA 15.0 for Week 52
Lobar pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 — MEDDRA 14.1 used for Week 26/MEDDRA 15.0 for Week 52
Cerebral infarction (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 — MEDDRA 14.1 used for Week 26/MEDDRA 15.0 for Week 52
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 — MEDDRA 14.1 used for Week 26/MEDDRA 15.0 for Week 52
Neophrolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 — MEDDRA 14.1 used for Week 26/MEDDRA 15.0 for Week 52
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 — MEDDRA 14.1 used for Week 26/MEDDRA 15.0 for Week 52
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 — MEDDRA 14.1 used for Week 26/MEDDRA 15.0 for Week 52
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 — MEDDRA 14.1 used for Week 26/MEDDRA 15.0 for Week 52
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 — MEDDRA 14.1 used for Week 26/MEDDRA 15.0 for Week 52
Diabetic foot (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 1 | 1 | 1 — MEDDRA 14.1 used for Week 26/MEDDRA 15.0 for Week 52
Skin necrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 — MEDDRA 14.1 used for Week 26/MEDDRA 15.0 for Week 52
Campylobacter gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 — MEDDRA 14.1 used for Week 26/MEDDRA 15.0 for Week 52. In the Week 26 study report, this event was coded as "campylobacter intestinal infection"; it was subsequently re-coded in the Week 52 study report as "campylobacter gastroenteritis".
Diabetic complications (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 — MEDDRA 14.1 used for Week 26/MEDDRA 15.0 for Week 52
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo: Baseline to Week 26 (N=90) | Canagliflozin 100 mg: Baseline to Week 26 (N=90) | Canagliflozin 300 mg: Baseline to Week 26 (N=89) | Placebo: Baseline to Week 52 (N=90) | Canagliflozin 100 mg: Baseline to Week 52 (N=90) | Canagliflozin 300 mg: Baseline to Week 52 (N=89)
Diarrhoea (Gastrointestinal disorders) | 5 | 3 | 4 | 9 | 4 | 4 — MEDDRA 14.1 used for Week 26/MEDDRA 15.0 for Week 52
Nasopharyngitis (Infections and infestations) | 10 | 3 | 7 | 13 | 5 | 9 — MEDDRA 14.1 used for Week 26/MEDDRA 15.0 for Week 52
Urinary tract infection (Infections and infestations) | 5 | 4 | 7 | 6 | 4 | 12 — MEDDRA 14.1 used for Week 26/MEDDRA 15.0 for Week 52
Hypoglycaemia (Metabolism and nutrition disorders) | 4 | 13 | 10 | 4 | 18 | 20 — MEDDRA 14.1 used for Week 26/MEDDRA 15.0 for Week 52
Vitamin D deficiency (Metabolism and nutrition disorders) | 5 | 0 | 1 | 4 | 2 | 1 — MEDDRA 14.1 used for Week 26/MEDDRA 15.0 for Week 52. In the Week 26 study report, 1 patient (placebo) had vitamin D deficiency recorded in error by the investigator which was corrected in the Week 52 study report.
Back pain (Musculoskeletal and connective tissue disorders) | 5 | 0 | 2 | 5 | 1 | 4 — MEDDRA 14.1 used for Week 26/MEDDRA 15.0 for Week 52
Dizziness (Nervous system disorders) | 0 | 1 | 5 | 2 | 1 | 5 — MEDDRA 14.1 used for Week 26/MEDDRA 15.0 for Week 52
Hypotension (Vascular disorders) | 0 | 1 | 6 | 3 | 1 | 6 — MEDDRA 14.1 used for Week 26/MEDDRA 15.0 for Week 52
Fatigue (General disorders) | 4 | 0 | 4 | 5 | 1 | 5 — MEDDRA 14.1 used for Week 26/MEDDRA 15.0 for Week 52
Oedema peripheral (General disorders) | 4 | 2 | 3 | 6 | 5 | 6 — MEDDRA 14.1 used for Week 26/MEDDRA 15.0 for Week 52
Bronchitis (Infections and infestations) | 3 | 4 | 3 | 1 | 5 | 5 — MEDDRA 14.1 used for Week 26/MEDDRA 15.0 for Week 52. Events for 2 patients in the placebo group in the Week 26 study report were reassessed as "chronic bronchitis" in the Week 52 study report.
Influenza (Infections and infestations) | 3 | 3 | 2 | 6 | 3 | 3 — MEDDRA 14.1 used for Week 26/MEDDRA 15.0 for Week 52
Upper respiratory tract (Infections and infestations) | 1 | 3 | 1 | 1 | 5 | 4 — MEDDRA 14.1 used for Week 26/MEDDRA 15.0 for Week 52
Hyperkalaemia (Metabolism and nutrition disorders) | 3 | 2 | 1 | 5 | 3 | 1 — MEDDRA 14.1 used for Week 26/MEDDRA 15.0 for Week 52
Hyperglycaemia (Metabolism and nutrition disorders) | 4 | 2 | 2 | 5 | 2 | 2 — MEDDRA 14.1 used for Week 26/MEDDRA 15.0 for Week 52
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 4 | 2 | 3 | 5 | 3 — MEDDRA 14.1 used for Week 26/MEDDRA 15.0 for Week 52
Headache (Nervous system disorders) | 3 | 2 | 2 | 5 | 3 | 3 — MEDDRA 14.1 used for Week 26/MEDDRA 15.0 for Week 52

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested in writing, such publication will be withheld for up to an additional 60 days.